CLINICAL TRIAL: NCT06933108
Title: Estimate the Risk of Diabetic and Uremic Peripheral Neuropathy Using Physical and Functional Testing
Brief Title: Prediction of Peripheral Neuropathy With Functional Testing
Acronym: PredictNP
Status: Recruiting | Type: Observational
Sponsor: Université catholique de l'Ouest (Other)
Collaborators: Centre Hospitalier le Mans (Other); Le Mans Universite (Other)
Responsible Party: Sponsor
Other Study IDs: UCO20250326
Record Dates: First submitted 2025-03-26; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Stage 3 and 4; Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Diabetes and chronic kidney disease (CKD) are two distinct pathologies. The former is defined as an impairment in insulin production and/or utilization, while the latter refers to structural or functional abnormalities of the kidneys. However, these two diseases share a common complication: peripheral neuropathy. This condition affects between 50% and 60% of patients with diabetes or CKD.

Peripheral neuropathy involves the destruction of sensory and motor neurons, leading to a wide range of painful symptoms while also reducing force production capacity. Among the diagnostic tests used, the most accessible clinical tests suffer from high variability due to human subjectivity (e.g., the tuning fork test, which requires examiner expertise and verbal patient feedback), whereas laboratory electrophysiological tests can only detect the largest neurons, which are affected at later stages. Although composite clinical tests have been developed to improve neuropathy screening performance, they still inherit the limitations of their individual components. In other words, they remain subject to variability related to the examiner's experience and the patient's ability to understand instructions, while also being performed through various procedures that lack a standardized consensus. Moreover, these composite scores are particularly time-consuming and are therefore rarely used in clinical practice. As a result, no method currently allows for large-scale, early, and reliable screening of peripheral neuropathy.

Our recent work and emerging studies suggest that assessing functional capacities could serve as an objective and early marker of neuropathic impairment, even before clinical diagnosis. Specifically, the quantification of postural balance performance using stabilometric methods (i.e., center of pressure displacement area) and unipedal balance time could predict the presence of diabetes-related peripheral neuropathy with over 95% accuracy compared to diagnosis with a composite clinical method (unpublished results).

Therefore, the aim of this study is to evaluate physical and balance capacities assessed during routine care in adapted physical activity settings, in order to determine whether the development of a composite score could help estimate the risk of peripheral neuropathy in individuals with diabetes and CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4-5 and / or diabetes (Type I or II)
* Able to walk 20 m
* BMI < 35

Exclusion Criteria:

* Currently or planning dialysis
* Musculoskeletal, osteorarticular and neurological disease(s)
* Cognitive impairment
* Low-limb amputation

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Le Mans Hospital, from nephrology and endocrinology unit
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Composite score derived from the statistical model | Transversal study : At baseline
  The composite score will be built with the performances at the functional tests (independant variables) using a logistic backward regression model, to predict peripheral neuropathy (dependant variable: yes or no). The score will range from 0 to 1. Higher is the score, higher is the risk of peripheral neuropathy.
  Dependant variables: Michigan Neuropathy Screening Instrument, to diagnosis peripheral neuropathy.
  Independant variables: Maximal dorsiflexion and plantar flexion of the ankle, maximal hallux flexion, 10-meter walking test (speed, cadence), postural balance, Timed-up and Go, and two proprioceptive tests (Joint Position Sense and the Star Excursion Balance Test).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: Undecided
Because the power of the prediciton will be based on the data. So the data cannot be shared before publication.